CLINICAL TRIAL: NCT00208988
Title: A Randomized Controlled Trial to Promote Physician-Patient Discussion of Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: 511-2005
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Prostate Cancer
Keywords: Health literacy; Physician-Patient Relationship; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: Educational handout about prostate cancer screening
Procedure: Simple cue for patient to talk to doctor

SUMMARY:
Prostate cancer is the most common type of cancer among men. It is also the second leading cause of cancer-related death among men. Two screening tests are available to try to detect prostate cancer early - the digital rectal examination (DRE) and the prostate specific antigen (PSA) blood test. Unfortunately, physicians aren't sure whether or not these two screening tests help save lives, and there's a lot of controversy about how to use them. Recently, a major government committee (the U.S. Preventive Services Task Force) recommended that physicians discuss the risks and potential benefits of prostate cancer screening with their patients, and allow patients to make their own decision.

Because of the controversies, many physicians currently don't discuss prostate cancer with their patients. The problem is that it takes time and effort to have these discussions, and the information is complicated. A lot of patients have trouble understanding it, especially if they have a limited educational background or trouble reading. When patients have difficulty obtaining, understanding, and acting on basic health information, we say that they have "low health literacy." Other researchers have shown that patients with low health literacy don't know as much about cancer screening and are less likely to get screened for various cancers. They also tend to be timid about discussing things with their doctor, and often go along with what the doctor says, rather than taking an active role in the decision making.

In 2003, under IRB approval, we conducted a study with 2 goals: 1) to encourage patients to talk to their doctor about prostate cancer screening, and 2) to learn more about the impact of low health literacy on these conversations. To promote conversation, we used two handouts, given to patients in the waiting room before they saw the doctor. The first was a patient education handout about prostate cancer screening, written in very simple terms with useful illustrations. The second was a handout that simply encouraged patients to talk to their doctor about prostate cancer. Patients got one of the two handouts, or a nutritional handout that served as a control. After they saw their doctor, a research assistant briefly interviewed the patient to find out whether or not prostate cancer screening was discussed. We also measured the patients' health literacy skills, and asked a few other questions about their decision to get screened for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 45-70

Exclusion Criteria:

* Unable to communicate in English
* Too ill
* In police custody
* Visual acuity worse than 20/60
* History of prostate cancer
* Lack of cooperation
* Overt psychiatric illnesses

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2003-05; Study Completion 2003-08

PRIMARY OUTCOMES:
Discussion of Prostate Cancer Screening

SECONDARY OUTCOMES:
DRE
PSA

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Kripalani, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Kripalani S, Sharma J, Justice E, Justice J, Spiker C, Laufman LE, Price M, Weinberg AD, Jacobson TA. Low-literacy interventions to promote discussion of prostate cancer: a randomized controlled trial. Am J Prev Med. 2007 Aug;33(2):83-90. doi: 10.1016/j.amepre.2007.03.018. PMID 17673094